CLINICAL TRIAL: NCT06150144
Title: The Efficacy and Safety of Using Intralesional 5-fluorouracil for Basal Cell Carcinoma: Clinical Trail
Brief Title: The Efficacy and Safety of Using Intralesional 5-fluorouracil for Basal Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aleppo (Other)
Collaborators: Aleppo University Hospital (Unknown)
Responsible Party: Principal Investigator, Ibrahim Arnaout, Principal Investigator, University of Aleppo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: intralesional 5-FU for BCC
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Basal Cell Carcinoma; BCC
Keywords: Surgical excision; Basal cell carcinoma; clinical Trail; intralesional 5-fluorouracil
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Fluorouracil; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with intralesional 5-fluorouracil. (Experimental)
  Interventions: Drug: 5-Fluorouracil
- Patients with Surgery (Active Comparator)
  Interventions: Other: SURGERY

INTERVENTIONS:
Drug: 5-Fluorouracil — The invistigators want to assess the safety and efficacy of using intralesional 5-FU for the management of different types of BCC (including all the types EXCEPT the infiltrative one), by estimating different outcomes after the intralesional administration of 5-FU to BCC patient. Patients are randomly selected from the outpatient dermatologic clinic in the Aleppo University Hospital (AUH) over a period of 12 months and then these patients are followed up over another 12 months.
  Other Names: 5-FU
  Arms: Patients with intralesional 5-fluorouracil.
Other: SURGERY — Total excision of the lesion
  Arms: Patients with Surgery

SUMMARY:
The investigators want to assess the safety and efficacy of using intralesional 5-FU for the management of different types of BCC (including all the types EXCEPT the infiltrative one), by estimating different outcomes after the intralesional administration of 5-FU to BCC patient. Patients are randomly selected from the outpatient dermatologic clinic in the Aleppo University Hospital (AUH) over a period of 12 months and then these patients are followed up over another 12 months.

DETAILED DESCRIPTION:
Brief Description: The investigatorswant to assess the safety and efficacy of using intralesional 5-FU for the management of different types of BCC (including all the types EXCEPT the infiltrative one), by estimating different outcomes after the intralesional administration of 5-FU to BCC patient. Patients are randomly selected from the outpatient dermatologic clinic in the Aleppo University Hospital (AUH) over a period of 12 months and then these patients are followed up over another 12 months.

Detailed Description: Clinicians routinely consider surgical removal as the best and sometimes the only cost-effective treatment of Basal cell carcinoma, but several studies have discussed other promising treatment approaches for BCC including 5% 5-FU cream which is indicated for the treatment of superficial BCC, in addition many studies have investigated the efficacy of the combination of 5-FU with Imiquimode or cryoablation presenting promising results, however when searching the medical literature there was only few studies dealing with types other than superficial BCC, in addition intralesional administration of 5-FU alone was not thoroughly assessed so far even though there are some studies showing positive results suggesting 5-FU to be a cost-effective alternative to surgical excision, but as these papers are asking for further studies and stronger evidence the invistigators decided to conduct this study in accordance with the best recommendations reached by latest medical literature.

ELIGIBILITY:
Inclusion Criteria:

* 5 Years to 90 Years (Child, Adult, Older Adult).
* Volunteer to participate in study
* Superficial lesion
* Nodular lesion (x ≤ 1.5 cm) patients are seen at the outpatient Department or in the dermatology wards at Aleppo University Hospital (AUH) over 12 months' period.

Exclusion Criteria:

* Ulcerative.
* Nodular lesion (x ≥ 1.5 cm)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Histologic complete response rate | 1 - 2 months
  defined by absence of any tumor on the basis of histologic analysis of the excised specimen.

SECONDARY OUTCOMES:
Sides effect | 1 year
  The patient will be monitored and followed up for 365 days after the injection.

CONTACTS AND LOCATIONS:
Overall Officials: Noura Abdulrahman, M.D., Principal Investigator — Department of Dermatology and Venereology, Faculty of Medicine, University of Aleppo, Aleppo, Syria; Rama Haj mharram, M.D., Study Director — Department of Dermatology and Venereology, Faculty of Medicine, University of Aleppo, Aleppo, Syria; Ahmad Yamen Arnaout, M.D., Study Director — Faculty of Medicine, University of Aleppo, Aleppo, Syria.; Silva Ishkhanian, PhD, Study Director — Department of Dermatology and Venereology, Faculty of Medicine, University of Aleppo, Aleppo, Syria
Locations (1):
- Ibrahim Arnaout, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: No
Not available to other researcher